CLINICAL TRIAL: NCT00770484
Title: Effects of Exercise in Orthostatic Intolerance
Brief Title: Effect of Exercise in OI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 080722
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Orthostatic Intolerance; Postural Tachycardia Syndrome
Keywords: Exercise; Propanolol; Beta blockers
MeSH Terms: conditions — Orthostatic Intolerance; Postural Orthostatic Tachycardia Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol then placebo (Experimental): Active treatment
  Interventions: Drug: Propranolol then Placebo
- Placebo then propranolol (Placebo Comparator): Placebo Treatment
  Interventions: Drug: Placebo then Propranolol

INTERVENTIONS:
Drug: Propranolol then Placebo — Propanolol 20 mg, given orally within 1 hour prior to exercising
  Other Names: Active
  Arms: Propranolol then placebo
Drug: Placebo then Propranolol — Placebo, matching pill given orally within 1 hour prior to exercising
  Other Names: Inactive
  Arms: Placebo then propranolol

SUMMARY:
The main limitation patients with orthostatic intolerance (OI, or postural tachycardia syndrome, POTS) have to exercise is related to their increase in heart rate when standing. Main pharmacological treatment today is aimed at reducing heart rate with the use of betablockers (propanolol), this theoretically could also improve their exercise capacity; if their heart rate do not increase as much with the medication, they could exercise more. In addition, it has been suggested that in healthy volunteers subjected to head down tilt for 2 weeks (situation that produces a "simulated" transient POTS-like state) a single bout of intense exercise can improve orthostatic tolerance the day after exercising. The mechanisms involved in such response are not that clear but could be an increase in plasma volume already diminished in POTS patients. It seems likely that the same could be true for POTS patients.

The purpose of the present study are to pharmacologically improve the amount of exercise POTS patients can perform by reducing their baseline heart rate (specific aim 1) and to evaluate next day heart responses to an acute bout of intense exercise.

Therefore, the specific aims of this study are:

1. To test the hypothesis that lowering heart rate response with propanolol will result in an increase in exercise capacity.
2. To test the hypothesis that a single bout of exercise will result in an improvement in orthostatic tolerance the day after exercising.

DETAILED DESCRIPTION:
* Subjects will be studied twice, once after receiving placebo and in a second occasion after receiving propanolol.
* An exercise capacity test with estimation of maximal oxygen consumption (VO2 max) will be done within 1 hour of receiving a pill containing placebo and that will be in appearance identical to the one for propanolol. This test will be conducted on a stationary bicycle and the effort will be gradually increased while expired air is measured during exhaustive physical work. The test will last approximately 30 minutes and be conducted in Vanderbilt's Clinical Trial Center.
* The day before and the day after the exercise test subjects will be asked to collect urine for 12 hours each time and to keep a record of how much liquid they ingest.
* Posture study tests (measurements of heart rate and blood pressure taken while lying down and at intervals for up to 30 minutes while standing) will be done the day before and the day after the exercise test.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria of POTS (Raj, et al., 2005)
* Age between 18-65 years
* Male and female are eligible (although the majority of patients POTS are female).
* Able and willing to provide informed consent

Exclusion Criteria:

* Presence of medical conditions that can explain postural tachycardia (e.g., dehydration, medications)
* Pregnancy
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol.
* Patients who are bedridden or chair-ridden.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Gamboa A, Okamoto LE, Raj SR, Diedrich A, Shibao CA, Robertson D, Biaggioni I. Nitric oxide and regulation of heart rate in patients with postural tachycardia syndrome and healthy subjects. Hypertension. 2013 Feb;61(2):376-81. doi: 10.1161/HYPERTENSIONAHA.111.00203. Epub 2013 Jan 2. PMID 23283362

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propranolol Then Placebo | Placebo Then Propranolol
Started | 8 | 4
Completed | 7 | 4
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol Then Placebo | Placebo Then Propranolol | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31 (3) | 32 (2) | 32 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximal Oxygen Consumption Capacity (VO2 Max)
Time Frame: Over approximately 30 minutes, within 2 hours of receiving each intervention.
Measure: Mean (Standard Error); unit: mL/kg/min
Groups:
- Propranolol: Active treatment
  Propranolol then Placebo: Propanolol 20 mg, given orally within 1 hour prior to exercising
- Placebo: Placebo Treatment
  Placebo then Propranolol: Placebo, matching pill given orally within 1 hour prior to exercising
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 11 | 11
mL/kg/min | 27.6 (1) | 24.5 (0.7)

ADVERSE EVENTS:
Arm/Group | Propranolol Then Placebo | Placebo Then Propranolol
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No